CLINICAL TRIAL: NCT07236697
Title: Impact of Subclinical Hypothyroidism on Liver Enzymes and Lipid Profile
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shahd Ali Mohamed, resident, Assiut University
Other Study IDs: 04-2025-201491
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Subclinical Hypothyroidism
Keywords: subclinical hypothyroidism on liver enzymes and lipid profile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: liver enzymes — subclinical hypothyroidism on liver enzymes and lipid profile

SUMMARY:
the goal of the randomized controlled observational study is to observe the effect of subclinical hypothyroidism on liver enzymes and lipid profile

DETAILED DESCRIPTION:
Subclinical hypothyroidism (SCH) is a prevalent endocrine disorder defined by elevated levels of thyroid-stimulating hormone (TSH) with normal concentrations of free thyroxine (T4) [1]. Despite its often-asymptomatic nature, SCH has been increasingly recognized for its association with a variety of metabolic abnormalities, with lipid profile disturbances being particularly notable[2].

The thyroid gland is one of the primary endocrine glands in human body and is in charge of the hormones triiodothyronine (T3) and thyroxine (T4). These hormones influence hepatic functions by regulating all cells' baseline metabolic rates, including hepatocytes. Therefore, any thyroid condition may impair liver function[3] .

sub clinical hypothyroidism is indicated by a moderate rise in TSH levels (TSH > 4 mIU/l), along with normal thyroid hormone levels. Approximately 3% of the general population is affected by overt hypothyroidism. However, sub clinical hypothyroidism is found in 5-10% of the global population, as well as 8-10% of individuals aged over 65 years [4]. It should be noted that thyroid hormones have a crucial impact on multiple organs, especially the liver[5]. SCH is more common in women, the elderly, and individuals with a family history of diabetes and thyroid diseases (6, 7)SCH patients had significantly higher triglyceride (TG) levels (1.69 ± 1.9 vs. 1.45 ± 1.4) than the healthy population [8]. Another study by Sindhu and Vijay (9) suggested that SCH patients had more significant dyslipidemia than the euthyroid population, including total cholesterol(TC),very low-density lipoprotein cholesterol (VLDL-C), and low-density lipoprotein cholesterol (LDL-C).

Subclinical hypothyroidism (SCH) contributes to the progression of metabolic dysfunction-associated steatotic liver disease (MASLD) through several mechanisms [10-12]. One significant mechanism involves the activity of thyroid-stimulating hormone (TSH) on the cell membrane of hepatocytes, which disrupts triglyceride metabolism in the liver.

Additionally, atherogenic dyslipidemia is commonly observed in patients with hypothyroidism. The primary cause of hyperlipidemia associated with hypothyroidism is a decrease in cholesterol excretion and a significant rise in apoB lipoproteins. This is mainly due to insufficient breakdown and turnover of cholesterol, stemming from a reduction in the number of low-density lipoprotein (LDL) receptors present on the surface of hepatocytes

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years

  * For SCH group: Elevated TSH with normal FT4
  * For control group: Normal TSH and FT4 levels

Exclusion Criteria:

* • Evident hypothyroidism or hyperthyroidism

  * Diagnosed with diabetes mellitus
  * Chronic liver disease
  * Chronic kidney disease
  * Use of lipid-lowering or thyroid medications
  * Pregnancy
  * Alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: internal medicine department
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Impact of Subclinical Hypothyroidism on Liver Enzymes and Lipid Profile | Baseline
  1. Mean levels of liver enzymes (ALT, AST, GGT)
     • To determine whether there is a statistically significant difference in liver enzyme levels between individuals with subclinical hypothyroidism and euthyroid controls.
  2. Mean values of lipid profile components (Total Cholesterol, LDL-C, HDL-C, Triglycerides) • To assess whether subclinical hypothyroidism is associated with dyslipidemia compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Abbas Said, professor, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shan Z, Chen L, Lian X, Liu C, Shi B, Shi L, Tong N, Wang S, Weng J, Zhao J, Teng X, Yu X, Lai Y, Wang W, Li C, Mao J, Li Y, Fan C, Teng W. Iodine Status and Prevalence of Thyroid Disorders After Introduction of Mandatory Universal Salt Iodization for 16 Years in China: A Cross-Sectional Study in 10 Cities. Thyroid. 2016 Aug;26(8):1125-30. doi: 10.1089/thy.2015.0613. Epub 2016 Jul 22. PMID 27370068
- [Result] Mavromati M, Jornayvaz FR. Hypothyroidism-Associated Dyslipidemia: Potential Molecular Mechanisms Leading to NAFLD. Int J Mol Sci. 2021 Nov 26;22(23):12797. doi: 10.3390/ijms222312797. PMID 34884625
- See also: Unraveling the Role of Hypothyroidism in Non-alcoholic Fatty Liver Disease Pathogenesis: Correlations, Conflicts, and the Current Stand — https://pubmed.ncbi.nlm.nih.gov/34104598/